CLINICAL TRIAL: NCT07106255
Title: Task-oriented Training Intervention for Multiple Sclerosis Patients
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Marie Carmen Valenza, Principal Investigator, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 036-N-23
Record Dates: First submitted 2025-07-17; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Task-oriented training program (Experimental): Task-oriented training program
  Interventions: Other: Task-oriented training
- Standard medical care and leaflet fatigue management (Active Comparator)
  Interventions: Other: Standar medical care and leaflet fatigue management

INTERVENTIONS:
Other: Task-oriented training — Participants included in the experimental group will underwent an 8-week TOT intervention, administered twice weekly, with each session lasting 45 minutes.
  Within this framework, the intervention will comprise sessions involving meaningful and repetitive activities tailored to both the patient and their specific context. The occupations will be selected by each participant through the Canadian Occupational Performance Measure (COMP) tool in the initial assessment. The activities were randomly ordered and focused on the reconstruction of complete tasks. To support task segmentation, a range of custom-designed materials will be employed, alongside therapeutic tools and materials such as therapeutic putty, TheraBand, and others commonly used in physical rehabilitation interventions. Throughout the intervention, participants will receive positive reinforcement that will fade over the time to prevent unnecessary dependency.
  Arms: Task-oriented training program
Other: Standar medical care and leaflet fatigue management — Participants included in the control group will continue with their usual treatment and will receive a pamphlet containing information on fatigue management.
  Arms: Standard medical care and leaflet fatigue management

SUMMARY:
This study aims to evaluate the effectiveness of a Task-oriented program in improving functional performance and health outcomes in patients with Multiple Sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Multiple Sclerosis by a neurologist.
* Aged over 18 years old.
* Acceptance and signature of the informed consent.

Exclusion Criteria:

* A cognitive level or condition that did not allow completion of the evaluations.
* An exacerbation of MS during the previous 3 months.
* Presence of interfering musculoskeletal, neurological, orthopaedic, and/or rheumatic disorders affecting hand and/or finger mobility, including previous trauma or fracture of the upper extremity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Occupational Performance | Baseline and at 8 weeks at the end of the intervention, and through study completion, at 1, 3, 6, and 12 months post-intervention (an average of 1 year)
  The main variable in this study will be the Canadian Occupational Performance Measure (COPM). This tool measures the perception of problems related to the overall quality of performance, development and satisfaction with particular occupations.

SECONDARY OUTCOMES:
Fatigue | Baseline and at 8 weeks at the end of the intervention, and through study completion, at 1, 3, 6, and 12 months post-intervention (an average of 1 year)
  The level of fatigue will be assessed with the Modified Impact Fatigue Scale (MFIS) and the Fatigue Severity Scale (FSS). The MFIS consists of items from which a total score is obtained and for each subscale. Scores range from 0 to 36 with higher scores indicating a greater impact of fatigue on activities. The FSS consists of 9 items that are rated on a scale of 1 to 7. A higher score indicates a higher agreement with the statement presented in each item.

OTHER OUTCOMES:
Upper limb strengh | Baseline and at 8 weeks at the end of the intervention, and through study completion, at 1, 3, 6, and 12 months post-intervention (an average of 1 year)
  Upper limb strength will be assessed using the Arm Curl Test (ACT). The ACT consists of performing as many arm curls as possible in 30 seconds while seated in a chair.
Upper limb strengh 2 | Baseline and at 8 weeks at the end of the intervention, and through study completion, at 1, 3, 6, and 12 months post-intervention (an average of 1 year)
  Upper limb strength will be assessed using a hand and pinch dynamometer. The dynamometer and hand dynamometer measure grip and pinch strength respectively.
Motor speed | Baseline and at 8 weeks at the end of the intervention, and through study completion, at 1, 3, 6, and 12 months post-intervention (an average of 1 year)
  Motor speed will be assessed with the Finger Tapping Test (FTT). In this test, the number of finger taps the participant is able to perform in three attempts of 20 seconds each is counted.
Manual dexterity - 9HPT | Baseline and at 8 weeks at the end of the intervention, and through study completion, at 1, 3, 6, and 12 months post-intervention (an average of 1 year)
  Manual dexterity will be assessed using the Nine Hole Peg Test (9HPT). 9HPT requires the participant to place and then remove nine pegs, one at a time, into nine holes on a board as quickly as possible. The test is performed separately with each hand, and the time taken to complete the task is recorded. Shorter completion times indicate better manual dexterity.
Manual dexterity - Purdue | Baseline and at 8 weeks at the end of the intervention, and through study completion, at 1, 3, 6, and 12 months post-intervention (an average of 1 year)
  Manual dexterity will be assessed using the Purdue Pegboard Test.
  Purdue Pegboard Test involves placing as many pins as possible into holes on a board. It includes subtests for dominant and non-dominant hand, both hands simultaneously, and an assembly task. Higher scores reflect better dexterity.
Manual dexterity - CRT | Baseline and at 8 weeks at the end of the intervention, and through study completion, at 1, 3, 6, and 12 months post-intervention (an average of 1 year)
  Manual dexterity will be assessed using the Coin Rotation Test (CRT).
  CRT assesses the coordination and speed of the fingers by rotating a coin clockwise with three fingers of the hand (thumb, index and middle finger) as fast as possible.
Satisfaction and adherence with the intervention | Baseline and at 8 weeks at the end of the intervention, and through study completion, at 1, 3, 6, and 12 months post-intervention (an average of 1 year)
  Satisfaction and adherence with the intervention will be recorded with the Sport Injury Rehabilitation Adherence Scale (SIRAS). Although originally designed for sport settings, it has been used to assess adherence and satisfaction in chronic populations.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Health Sciences. University of Granada, Granada, Granada, Spain